CLINICAL TRIAL: NCT03949790
Title: Erector Spinae Plane Block Combined With Intercostal Nerve Block in Video Assisted Thoracoscopic Surgery: a Randomized Study
Brief Title: ESPB Combined With Intercostal Nerve Block in VATs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Tae Kyong Kim, Assistant Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2019-107
Record Dates: First submitted 2019-05-06; First posted 2019-05-14 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Video Assisted Thoracoscopic Surgery

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intercostal block with ESPB (Active Comparator): Performed ESPB in VATs with intercostal nerve block
  Interventions: Procedure: ESPB and Intercostal nerve block
- Intercostal block without ESPB (Active Comparator): Not Performed ESPB in VATs with intercostal nerve block
  Interventions: Procedure: Intercostal nerve block

INTERVENTIONS:
Procedure: ESPB and Intercostal nerve block — Erector spinae plane block + Intercostal nerve block
  Arms: Intercostal block with ESPB
Procedure: Intercostal nerve block — Intercostal nerve block
  Arms: Intercostal block without ESPB

SUMMARY:
A randomized prospective trial to test the effect of additional Erector Spinae Plane Block (ESPB) with intercostal nerve block during video assisted thoracoscopic surgery.

DETAILED DESCRIPTION:
A prospective randomized trial which aims to evaluate effect of peripheral nerve block for pain management, the Erector Spinae Plane Block (ESPB) in patients undergoing video assisted thoracoscopic surgery with intercostal nerve block.

ELIGIBILITY:
Inclusion Criteria:

* Wedge Resection or Lobectomy under VATS approach.

Exclusion Criteria:

* Age < 20 years
* Patients who has anatomical abnormality in any spine
* Patients who has skin infection near to be the present procedure site
* Intercostal nerve block is not performed during surgery
* Previous lung surgery history of affected side

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-06-18 (Actual); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-07-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative Pain | 1 hour after surgery
  VAS score (Visual Analog Scale for Pain, 0-10, higher value represent a worse outcome)

SECONDARY OUTCOMES:
Postoperative Pain | 6 hours after surgery
  VAS score (Visual Analog Scale for Pain, 0-10, higher value represent a worse outcome)
Postoperative Pain | 12 hours after surgery
  VAS score (Visual Analog Scale for Pain, 0-10, higher value represent a worse outcome)
Postoperative Pain | 24 hours after surgery
  VAS score (Visual Analog Scale for Pain, 0-10, higher value represent a worse outcome)
Postoperative Pain | 48 hours after surgery
  VAS score (Visual Analog Scale for Pain, 0-10, higher value represent a worse outcome)
Opioid consumption | postoperative 24 hours
  cumulative total opioid consumption

CONTACTS AND LOCATIONS:
Overall Officials: Tae Kyong Kim, MD, phD, Study Chair — SMG-SNU Boramae
Locations (1):
- SMG - SNU Boramae Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chin KJ, Adhikary S, Sarwani N, Forero M. The analgesic efficacy of pre-operative bilateral erector spinae plane (ESP) blocks in patients having ventral hernia repair. Anaesthesia. 2017 Apr;72(4):452-460. doi: 10.1111/anae.13814. Epub 2017 Feb 11. PMID 28188621
- [Background] Forero M, Rajarathinam M, Adhikary S, Chin KJ. Continuous Erector Spinae Plane Block for Rescue Analgesia in Thoracotomy After Epidural Failure: A Case Report. A A Case Rep. 2017 May 15;8(10):254-256. doi: 10.1213/XAA.0000000000000478. PMID 28252539
- [Background] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016
- [Background] Hamilton DL, Manickam B. Erector spinae plane block for pain relief in rib fractures. Br J Anaesth. 2017 Mar 1;118(3):474-475. doi: 10.1093/bja/aex013. No abstract available. PMID 28203765
- [Background] Forero M, Rajarathinam M, Adhikary S, Chin KJ. Erector spinae plane (ESP) block in the management of post thoracotomy pain syndrome: A case series. Scand J Pain. 2017 Oct;17:325-329. doi: 10.1016/j.sjpain.2017.08.013. Epub 2017 Sep 12. PMID 28919152